CLINICAL TRIAL: NCT01822197
Title: Pilot Trial of Phototherapy for Acute Depression in Hospitalized CF Patients
Brief Title: Pilot Trial of Phototherapy for Acute Depression in Hospitalized Cystic Fibrosis Patients
Acronym: PHOTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Kopp, Principal Investigator, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB13-00044
Record Dates: First submitted 2013-03-25; First posted 2013-04-02 (Estimated); Results first posted 2016-09-07 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-10

CONDITIONS: Depression; Cystic Fibrosis
Keywords: Phototherapy
MeSH Terms: conditions — Depression; Cystic Fibrosis | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phototherapy (Experimental): Bright light phototherapy will be administered for 30 minutes daily over one week in the morning (Days 0-7)
  Interventions: Device: Phototherapy

INTERVENTIONS:
Device: Phototherapy — light will be administered at a minimum distance of 12 inches away to provide 10,000 lux
  Other Names: Nature Bright Sun Touch Plus light box.

SUMMARY:
The purpose of this study is to determine whether bright light phototherapy can improve depressive symptoms in hospitalized patients with cystic fibrosis (CF) with subsequent effects on quality of life and illness recovery. It is hypothesized that phototherapy will improve depressive symptoms and decrease length of stay in depressed patients with CF who are hospitalized.

DETAILED DESCRIPTION:
Adults and adolescent with CF who are admitted to the hospital for pulmonary exacerbations will be enrolled. Subjects will use a Sun Touch Plus light box that emits 10,000 lux at a minimum distance of 60-80 cm away upon first awakening. Light exposure will last for 30 minutes each day over one week. Nursing staff will ensure compliance and a light sensor attached to the light box will measure use as well. There will not be a placebo during this pilot trial due to recruitment concerns for the sample size required for a single center placebo controlled trial. All light boxes will be sterilized between patient use. Vitamin D levels will be recorded at enrollment from routine clinical measurement. Light boxes do NOT emit UV light and have a negative ionizer.

Depression Screening: Quick Inventory of Depressive Symptomatology self report and clinician administered survey (QIDS-SR and QIDS-C) will be administered at admission (day 0) and completion of light therapy (day 7) to look at changes in depressive symptoms. The QIDS assesses all the criterion symptom domains designated by the American Psychiatry Association Diagnostic and Statistical Manual of Mental Disorders - 4th edition (DSM-IV) to diagnose a major depressive episode. The QIDS is sensitive to change, with medications, psychotherapy, or somatic treatments, making it useful for research purposes. The psychometric properties of both the QIDS has been established in various study samples. Cronbach's alpha was 0.85 (QIDS-C16) and 0.86 (QIDS-SR16) in a reliability study by Triveldi in 2004.

Quality of Life Scoring: The CF questionnaire revised (CFQ-R) will be administered simultaneously with the QIDS at days 0 & 7 as a measure of health related quality of life (HRQOL). This is a well validated measure in the CF population for research studies (Riekert et al., 2007).

ELIGIBILITY:
Inclusion Criteria:

* Patients with CF greater than 12 years of age
* Pulmonary exacerbation

Exclusion Criteria:

* planned admission less than 24 hours
* suicidal ideation
* Bipolar depression
* known retinal disorder/photosensitivity
* light induced epilepsy or migraines
* age less than 12 years of age

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin T Kopp, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phototherapy
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phototherapy
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (8.5)
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospitalization
Description: Length of stay will be measured in days
Time Frame: participants will be followed for the length of hospital stay, an average of 14 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phototherapy
Number analyzed (Participants) | 30
days | 11 (3.6)

2. Secondary Outcome: Depressive Symptom Scores Post-Treatment (Day 7) and at Admission (Day 0)
Description: depressive symptom scoring at day 0 and day 7 using Quick Inventory of Depressive Symptomatology-clinician (QIDS-C) and Quick Inventory of Depressive Symptomatology self-report (QIDS-SR). Day 7 and Day 0 scores will be compared. Score range is 0 to 27. A QIDS score of less than 6 indicates no depression, 6-10 indicates mild depression, 11-15 moderate, 16-20 severe, and 21- 27 very severe depression.
Time Frame: between day 0 and day 7 of hospitalization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phototherapy
Number analyzed (Participants) | 30
units on a scale
  Post-treatment score | 4.5 (2.5)
  Admission score | 8.7 (3.6)

3. Secondary Outcome: Quality of Life Scoring Post-Treatment (Day 7) and at Admission (Day 0
Description: Quality of life scoring at admission (Day 0) and post-treatment (Day 7) using the CF questionnaire-revised (CFQ-R) as a measure of health related quality of life. Minimally important changes in CFQ-R scoring have been reported at 5-8. Days 0 and 7 will be compared. Score range is 0 to 100. Lower scores indicate worse quality of life.
Time Frame: between day 0 and day 7 of hospitalization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phototherapy
Number analyzed (Participants) | 30
units on a scale
  Pre-treatment Health Domain | 35.5 (17.1)
  Post-treatment health domain | 59.7 (16.7)

ADVERSE EVENTS:
Arm/Group | Phototherapy
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No